CLINICAL TRIAL: NCT02834923
Title: Enhancing Self-Management Support in Diabetes Through Patient Engagement
Acronym: EE-CTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Colorado, Denver (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-17033; R18DK108039-05 (NIH)
Record Dates: First submitted 2016-07-06; First posted 2016-07-15 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Cystathionine gamma-Lyase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Connection to Health (CTH) (Active Comparator): CTH is a comprehensive SMS program that focuses on behavior change. CTH utilizes web-based interactive behavior change technology, based on a logic model of behavior and maintenance that is informed by social-cognitive and social ecological theories. Prior to diabetes visits with a clinician, health educator, or care manager, patients complete a pre-visit CTH assessment at their practice through a tablet computer or computer kiosk. CTH assesses multiple diabetes management behaviors (diet, physical activity, medication adherence, alcohol and tobacco use, stress, mood) using brief assessment measures, each with cut-points highlighting areas of deficit. Action planning plays a central role, through a web-based platform that allows the patient and health care team to select and set goals collaboratively.
  Interventions: Behavioral: Connection to Health (CTH)
- Enhanced Engagement Protocol for CTH (EE-CTH) (Experimental): EE-CTH seamlessly integrates CTH with an efficacious, structured, motivational interview (MI)-informed protocol specifically designed to enhance patient engagement in SMS activities. Key components of MI have been incorporated into a practical and systematic engagement protocol that includes: (1) acknowledging the patient's point of view; (2) identifying and labeling the patient's ambivalence (both the good reasons for making the change and the good reasons for not making the change); (3) evaluating whether change is really worth the effort; (4) identifying, reflecting and labeling accompanying feelings and concerns about change; and (5) establishing a small and meaningful goal by the end of the encounter.
  Interventions: Behavioral: Enhanced Engagement Protocol for CTH (EE-CTH)

INTERVENTIONS:
Behavioral: Enhanced Engagement Protocol for CTH (EE-CTH) — EE-CTH integrates CTH with an efficacious, structured, motivational interview (MI)-informed protocol.
  Arms: Enhanced Engagement Protocol for CTH (EE-CTH)
Behavioral: Connection to Health (CTH) — CTH is a comprehensive SMS program that focuses on behavior change.
  Arms: Connection to Health (CTH)

SUMMARY:
The Patient Centered Medical Home (PCMH) and the Chronic Care Model (CCM) are complementary clinical intervention frameworks that are commonly invoked to support better type 2 diabetes (T2DM) outcomes in primary care. Self-management Support (SMS) is a core component of both the PCMH and CCM, and focuses on the central role of patients in managing their illness by engaging with and adopting healthy behaviors that promote optimal clinical outcomes. Despite its recognized importance, SMS programs for diabetes continue to demonstrate limited effectiveness in the real-world of primary care.

SMS is comprised of two complementary and interactive components: (1) patient engagement (e.g., the process of eliciting and responding to patients emotions and motivations related to health behaviors), and (2) behavioral change tools (e.g., selecting specific goals, creating action plans). While several sophisticated SMS programs have been developed for T2DM, the vast majority are designed with a narrow focus on behavioral change tools, largely ignoring unique aspects of the patient context that drive and maintain health behavior. Considerable clinical research suggests that the addition of a structured, evidenced-based program of patient engagement can maximize the effectiveness of SMS programs for patients with T2DM in primary care.

To date there has been no systematic study of the degree to which fully integrating enhanced patient engagement as part of SMS will increase the initiation and maintenance of behavior change over time, and for which kinds of patients enhanced patient engagement is essential. To address this gap, the investigators will compare a state-of-the-art, evidence-based SMS behavior change tool program, called Connection to Health (CTH), with an enhanced CTH program that includes a practical, time-efficient patient engagement protocol, to create a program with an integrated and comprehensive approach to SMS, called "Enhanced Engagement CTH" (EE-CTH). The current study will directly test the added benefit of EE-CTH to CTH with regard to self-management behaviors and glycemic control in resource-limited community health centers, where vast numbers of patients with T2DM from ethnically diverse and medically vulnerable populations receive their care. The investigators will use an effectiveness-implementation hybrid design, employing the "Reach Effectiveness Adoption Implementation Maintenance" (RE-AIM) framework to test these two SMS programs for T2DM. This will provide critical information that will support dissemination and implementation of effective SMS programs in resource-limited primary care settings, serving diverse and medically vulnerable populations with much to gain from improved SMS.

DETAILED DESCRIPTION:
This is a two-arm, 14 month pragmatic cluster randomized trial to evaluate the added benefit of EE-CTH relative to CTH for patients with T2DM in primary care.

Primary care practices (not patients) will be randomly assigned to receive and deliver CTH or EE-CTH in an innovative effectiveness-implementation hybrid design. Using the RE-AIM framework, the investigators will evaluate program effectiveness in a real world setting, while at the same time gathering information on program reach, adoption, implementation and maintenance. CTH and EE-CTH practice trainings and delivery will each follow separate and standardized protocols, with support provided to practices through staff training, ongoing supervision and case presentations, and a practice improvement team assisted by a practice facilitator to address issues of staffing and patient flow. Practice training and facilitation notes, in conjunction with feedback from patient advisory councils, will be captured and integrated to identify barriers and facilitators to the implementation process and inform dissemination efforts. Beyond the requirements of the study, practices will be permitted to use EE-CTH or CTH with other patients as wished, which will enable the investigators to document the program's reach within the practice. Patients in both study arms will receive the intervention at a minimum of two primary care appointments (baseline and follow-up between 6 and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes;
* Diagnosed and receiving care at participating practices for at least 12 months;
* Able to read in English or Spanish (at least 6th grade level).

Exclusion Criteria:

* Not meeting all inclusion criteria

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 725 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycated haemoglobin) | Change from baseline to follow-up (6 to 12 months)
  Percentage HbA1c
High fat food | Change from baseline to follow-up (6 to 12 months)
  Amount of high fat food consumed weekly adapted from the Summary of Diabetes Self-Care Activities
Physical activity | Change from baseline to follow-up (6 to 12 months)
  Number of minutes of participation in physical activity from the International Physical Activity Questionnaire
Number of days missed medications | Change from baseline to follow-up (6 to 12 months)
  Number of days missed missing one or more medications in the past 14 days
Medication adherence | Change from baseline to follow-up (6 to 12 months)
  Frequency of reasons for missing medications.
Fruit and vegetable intake | Change from baseline to follow-up (6 to 12 months)
  Number of daily fruit and vegetable servings adapted from the Summary of Diabetes Self-Care Activities
Sugar-sweetened beverages | Change from baseline to follow-up (6 to 12 months)
  Number of daily sugar-sweetened beverages from the Starting the Conversation Measure

SECONDARY OUTCOMES:
Health-related distress | Change from baseline to follow-up (6 to 12 months)
  Modified from the Diabetes Distress Scale
Depression symptoms | Change from baseline to follow-up (6 to 12 months)
  Patient Health Questionnaire (PHQ8) Score
Weight | Change from baseline to follow-up (6 to 12 months)
  Weight (pounds)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Hessler, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Fisher L, Glasgow RE, Mullan JT, Skaff MM, Polonsky WH. Development of a brief diabetes distress screening instrument. Ann Fam Med. 2008 May-Jun;6(3):246-52. doi: 10.1370/afm.842. PMID 18474888
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Background] Paxton AE, Strycker LA, Toobert DJ, Ammerman AS, Glasgow RE. Starting the conversation performance of a brief dietary assessment and intervention tool for health professionals. Am J Prev Med. 2011 Jan;40(1):67-71. doi: 10.1016/j.amepre.2010.10.009. PMID 21146770
- [Derived] Hessler D, Fisher L, Dickinson M, Dickinson P, Parra J, Potter MB. The impact of enhancing self-management support for diabetes in Community Health Centers through patient engagement and relationship building: a primary care pragmatic cluster-randomized trial. Transl Behav Med. 2022 Oct 7;12(9):909-918. doi: 10.1093/tbm/ibac046. PMID 36205473